CLINICAL TRIAL: NCT07078513
Title: Active Release Technique Versus Strain-Counter Strain in Improving Pain and Function in Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01016 Asad Zaman
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Plantar Fascitis
Keywords: Plantar fasciitis; Chronic Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active release Technique (Experimental): Participants in this group will receive Active Release Technique (ART), a manual therapy approach focused on relieving soft tissue restrictions. The therapist will apply targeted pressure to areas of adhesion while the patient actively moves the affected tissue through its full range of motion. Each session will include approximately 30 repetitions and will be conducted three times per week for four weeks. This technique aims to restore normal tissue mobility and reduce pain.
  Interventions: Other: Active release Technique
- Strain counter strain tecnhnique (Experimental): Participants in this group will receive Strain-Counterstrain (SCS), a gentle manual therapy technique designed to reduce muscle tension and pain. The therapist will passively position the patient into a position of maximal comfort, targeting specific tender points. This position is held for approximately 90 seconds while maintaining light pressure, allowing the muscle and fascia to relax. Sessions will be conducted three times per week for four weeks, aiming to restore tissue balance and reduce discomfort.
  Interventions: Other: Strain counter strain tecnhnique

INTERVENTIONS:
Other: Active release Technique — Active Release Technique (ART) is a hands-on manual therapy that targets soft tissue restrictions by combining precise pressure with patient-assisted movement. It helps break down adhesions, improve mobility, and reduce pain by restoring normal tissue function.
  Arms: Active release Technique
Other: Strain counter strain tecnhnique — Strain-Counterstrain is a gentle, passive manual therapy that relieves muscle tension by positioning the body in a pain-free, comfortable posture. The therapist holds this position for about 90 seconds while applying light pressure to tender points, allowing the muscle and fascia to relax and reset.
  Arms: Strain counter strain tecnhnique

SUMMARY:
This randomized controlled trial compares the effectiveness of Active Release Technique (ART) and Strain-Counterstrain (SCS) in treating plantar fasciitis. Forty participants will be divided into two groups receiving either ART or SCS over a four-week period. The study aims to identify the more effective manual therapy technique for reducing pain and improving function in patients with plantar fasciitis.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the comparative effectiveness of Active Release Technique (ART) and Strain-Counterstrain (SCS) in managing plantar fasciitis, a common cause of heel pain and functional limitation. Forty participants will be randomly assigned to two intervention groups, each receiving either ART or SCS over a four-week period, with sessions conducted three times per week. ART involves targeted pressure with active tissue movement to release adhesions, while SCS uses passive positioning to relieve muscle tension. The study will be conducted at Bacha Khan Medical Complex, Swabi. Data will be analyzed using appropriate statistical methods to determine the superior technique. The findings aim to support evidence-based manual therapy approaches in clinical physiotherapy practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 25-45 years diagnosed with plantar fasciitis.
* Chronic plantar fasciitis (symptoms lasting more than 3 months).
* Ability to participate in active movement for ART.

Exclusion Criteria:

* Recent lower limb surgery.
* Neurological disorders affecting gait or mobility.
* Acute inflammatory conditions of the foot.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
NPRS | four weeks
  The Numeric Pain Rating Scale (NPRS) is a 0 to 10 self-reported scale used to assess pain intensity, where 0 = no pain and 10 = worst possible pain. It is a simple, reliable tool commonly used in clinical trials to measure pain levels before and after interventions.
Foot Function Index (FFI) | Four weeks
  Functional mobility will be assessed using the Foot Function Index (FFI), a validated self-reported questionnaire designed to measure the impact of foot pathology on pain, disability, and activity limitation in daily life.
Goniometer | Four weeks
  a reliable and widely used clinical tool that measures joint angles in degrees. It helps quantify movement limitations and improvements in specific planes, such as flexion, extension, abduction, and rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Zavata Afnan, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Chakdara, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No